CLINICAL TRIAL: NCT06054529
Title: Spatiotemporal Dimensions of Metabolism in Autochthonous Tumors of GBM Patients
Acronym: GBM-FLUX2
Status: Active, not recruiting | Type: Observational
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2063291
Record Dates: First submitted 2023-09-20; First posted 2023-09-26 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Niacinamide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants in surgery: Surgical removal of the GBM tumor.
  Interventions: Procedure: Surgical removal of the GBM tumor; Other: d4-NAM infusion

INTERVENTIONS:
Procedure: Surgical removal of the GBM tumor — Surgical removal of the GBM tumor
Other: d4-NAM infusion — Following the surgical removal of the GBM tumor, GBM patients will be dosed with a form of nicotinamide (a natural vitamin) that we can track. The nicotinamide will be converted to methyl nicotinamide (MeNAM) in the tumor. We will measure how fast the nicotinamide is converted to methyl nicotinamide. We believe that the speed of this chemical reaction in the tumor (fast versus slow) may be correlated with GBM aggressiveness.
  Other Names: Nicotinamide

SUMMARY:
To learn how altered metabolism in GBM causes tumor growth and resistance to drug therapy. In this pilot research study, we will dose GBM patients with a form of nicotinamide (a natural vitamin) that we can track. The nicotinamide will be converted to methyl nicotinamide (MeNAM) in the tumor. We will measure how fast the nicotinamide is converted to methyl nicotinamide. We believe that the speed of this chemical reaction in the tumor (fast versus slow) may be correlated with GBM aggressiveness

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative MRI consistent with a primary intracranial malignant brain tumor.
2. Must be 18 years of age or older.
3. Patient eligible for debulking surgery/resection.

Exclusion Criteria:

1. Inability to obtain pre-operative IV access.
2. Use of Tru Niagen, Basis (or any other nicotinamide riboside (NR)-containing NAD+ booster) or niacin supplements within one month prior to Study Visit 1.
3. Participation in studies involving investigational drug(s) within 30 days prior to Study Visit 1
4. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to Study Visit 1 (participants may not donate blood any time during the study, through the final study day)
5. Presence of any condition that, in the opinion of Dr. Field, compromises participant safety or data integrity or the participant's ability to complete study days.
6. Pregnancy, lactation or < 9 months postpartum from the Study Visit 1 date.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The research being pursued in this study is relevant to all GBM patients including these who are cognitively impaired.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Subtyping of GBM tumors as Classical, Proneural or MES (based on RNA-seq) | 2 months
  Resected tumor tissue will undergo routine testing

CONTACTS AND LOCATIONS:
Overall Officials: Adeline Divoux, PhD, Principal Investigator — AdventHealth Translational Research Institute
Locations (1):
- AdventHealth Translational Research Institute, Orlando, Florida, United States